CLINICAL TRIAL: NCT03006601
Title: Effect of Vision Therapy on Accommodation in Myopic Chinese Children With Poor Accommodative Response: A Randomized Clinical Trial
Brief Title: Effect of Vision Therapy in Myopic Children With Poor Accommodative Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiang Chen, Study Principal Investigator Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016AC2
Record Dates: First submitted 2016-10-28; First posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo group (Placebo Comparator): After enrollment, patients will be randomized into either treatment group or placebo group. Patients will receive placebo procedure which were designed to look like real vergence/accommodative therapy procedures yet not stimulate vergence, accommodation, of fine saccadic eye movement skills beyond normal daily visual activities. Office-based procedures (60 minutes per visit, one time per week, 12 weeks) and home procedures (15 minutes each time, five times per week, 12 weeks) will be provided to patients.
  Interventions: Other: Office-based accommodative/vergence therapy
- Treatment group (Experimental): After enrollment, patients will be randomized into either treatment group or placebo group. Office-based accommodative/vergence therapy (60 minutes per visit, one time per week, 12 weeks) and home reinforcement (15 minutes each time, five times per week, 12 weeks) will be provided to patients of treatment group.
  Interventions: Other: Office-based accommodative/vergence therapy

INTERVENTIONS:
Other: Office-based accommodative/vergence therapy — Office-based accommodative/vergence therapy (60 minutes per visit, one time per week, 12 weeks) and home reinforcement (15 minutes each time, five times per week, 12 weeks)

SUMMARY:
This study aims to determine the treatment effect of vision therapy on myopic children by assessment of accommodative function before and after therapy.

DETAILED DESCRIPTION:
1. Specific aims of the proposed clinical trial:

   1.1 To provide a definitive proof that vision therapy (VT) can improve the accommodative function of myopic children by comparing the results from treatment group to placebo group.

   1.2 To minimize the influences of confounding variables by randomly assigning the intervention.

   1.3 To observe the longitudinal effects of VT on accommodation system and its effect on axial length.
2. Hypothesis:

VT can improve the accommodative functions of 8-12 years old Chinese myopic children with poor accommodative response.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in the trial must:

* be within the age range of 8 to 12 years old inclusive
* -0.75D to -4.50Dspherical equivalent by cycloplegic autorefraction in both eyes
* astigmatism≤1.5D in both eyes
* anisometropia≤1.0D
* monocular accommodation lag at near(33cm)in right eye by non-cycloplegic autorefraction≧1D
* have vision correctable to at least 0.8 or better in each eye.

Exclusion Criteria:

Subjects enrolled in the trial must NOT have:

* current or prior use of PALs, bifocals, or contact lenses in either eye( prior or current use of SVLs allowed)
* history of any of the following functional defects: strabismus, amblyopia, nystagmus
* history of diabetes or seizures
* history of any ocular systemic, or neuro-developmental condition that might influence refractive development
* use of ocular or systemic medications containing atropine, pirenzepine, and anti-epileptic medications in recent 3 months
* history of any ocular surgery that might influence refractive development
* developmental disability, attention deficit hyperactivity disorder(ADHD), or learning disability diagnosis in children that in the investigator's discretion would interfere with office-based treatment
* relocation anticipated for 1 year
* birth weight lower than 1250 grams（2lbs,12oz）
* siblings in the study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2016-09; Primary Completion 2017-02 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the change of Accommodative response is being assessed | At least 15 visits (Screening visit, baseline visit, 12 weekly visits and 6 months after therapy). Eye examination will only be performed at screening visit, baseline visit, 6 week follow up, 12 week follow up,6 months after VT.
  we will use objective measures from open-field auto refractor.

SECONDARY OUTCOMES:
the changes of Accommodative amplitude is being assessed: | At least 15 visits (Screening visit, baseline visit, 12 weekly visits and 6 months after therapy). Eye examination will only be performed at screening visit, baseline visit, 6 week follow up, 12 week follow up,6 months after VT.
  we will use subjective measures from accommodative rod(push up method)
the changes of Accommodative facility is being assessed: | At least 15 visits (Screening visit, baseline visit, 12 weekly visits and 6 months after therapy). Eye examination will only be performed at screening visit, baseline visit, 6 week follow up, 12 week follow up,6 months after VT.
  we will use subjective measures from lens flipper
the changes of Cycloplegic objective refraction is being assessed: | At least 15 visits (Screening visit, baseline visit, 12 weekly visits and 6 months after therapy). Eye examination will only be performed at screening visit, baseline visit, 6 week follow up, 12 week follow up,6 months after VT.
  we will use objective measures from open-field auto refractor.
the changes of Axial length is being assessed: | At least 15 visits (Screening visit, baseline visit, 12 weekly visits and 6 months after therapy). Eye examination will only be performed at screening visit, baseline visit, 6 week follow up, 12 week follow up,6 months after VT.
  we will use objective measures from IOL-Master

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Chen, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided